CLINICAL TRIAL: NCT05365087
Title: The Effect of Endoscopic Fundoplication Prior to Sleeve Gastrectomy Versus Gastric Bypass on Reflux Symptoms in Bariatric Patients With Gastroesophageal Reflux Disease
Brief Title: Transoral Fundoplication Prior to Sleeve Gastrectomy Versus RNY Gastric Bypass on GERD Symptoms in Bariatric Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Lexington Health Incorporated (Other)
Responsible Party: Principal Investigator, Marc Antonetti, MD, Principal Investigator, Lexington Health Incorporated
Other Study IDs: LMC2021-1001
Record Dates: First submitted 2022-04-04; First posted 2022-05-09 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-03

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Gastric Bypass

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- TS Cohort: Patients who chose the Transoral Fundoplication TF prior to the Laparoscopic Sleeve Gastrectomy LSG procedure.
  Interventions: Procedure: Transoral Fundoplication and Sleeve Gastrectomy
- RNY Cohort: Patients who chose the Laparoscopic Roux-enY Gastric Bypass procedure.
  Interventions: Procedure: Gastric Bypass
- LSG Cohort: Patients with no evidence of GERD who undergo LSG and complete standard surveillance endoscopy

INTERVENTIONS:
Procedure: Transoral Fundoplication and Sleeve Gastrectomy — Transoral Fundoplication procedure completed prior to Sleeve Gastrectomy
  Groups: TS Cohort
Procedure: Gastric Bypass — Laparoscopic Roux-en-Y gastric bypass
  Groups: RNY Cohort

SUMMARY:
A retrospective and prospective cohort study to compare the effect of completing a Transoral Fundoplication procedure prior to Laparoscopic Sleeve Gastrectomy surgery to Laparoscopic Roux-en-Y Gastric Bypass in bariatric patients with Gastroesophageal Reflux Disease signs and symptoms. The aim of this study is to examine the effect of TF prior to sleeve gastrectomy as compared to Roux-en-Y Gastric Bypass on reflux symptoms in bariatric patients. Additional Follow up data until 10 years will be collected to evaluate for sequelae of GERD.

DETAILED DESCRIPTION:
Gastroesophageal Reflux Disease or GERD is a common condition that produces discomfort and can result in serious sequelae from frequent esophageal acid exposure, including Barrett's esophagus, erosive esophagitis, esophageal adenocarcinoma, voice changes, and asthma exacerbation. The prevalence of GERD in adults continues to increase in conjunction with the increase in obesity. Because obesity and GERD are clearly linked, an individual with obesity is four times more likely to develop esophageal carcinoma than in an individual with a normal BMI. Additionally, the incidence of GERD is proportional to rising BMI ranging from 23 to 50%. Weight loss is associated with decreased GERD symptoms. Bariatric surgery has proven to be effective in reducing BMI, which subsequently often reduces GERD. The laparoscopic sleeve gastrectomy is an effective weight loss tool; however, recent literature suggests a correlation of de novo or worsening reflux symptoms in bariatric patients within one year postoperatively, independent of weight loss. A study conducted by Tai,et al,.2013 found that the prevalence of GERD symptoms increased significantly from 12.1% to 47% after LSG. Additionally, of the 58 patients in the study who were asymptomatic prior to surgery, 44.8% developed GERD symptoms after LSG. Other studies have found that among patients with no preoperative GERD, 86% developed symptoms postoperatively.

The Laparoscopic Roux-en-Y gastric bypass has been touted as the gold standard to treat both obesity and GERD; however, this procedure has a higher morbidity rate. While LSG has relatively low rates of re-operations, the LRYGB carries significant lifetime risk for multiple operative procedures due to adhesive bowel obstruction, internal hernia, non-healing ulcers and intussusception. Furthermore, nutrient malabsorption following LRYGB can result in irreversible neurological complications, and accelerated, ongoing decline in bone mineral density.. Options for surgical correction of GERD are limited following bariatric surgery. However, options for anti-reflux procedures prior to undergoing bariatric surgery are viable, and may include Transoral Fundoplication.

Transoral fundoplication is an anti-reflux procedure which has proven to achieve long-lasting relief of gastroesophageal reflux symptoms, and eliminate, or reduce the use of proton pump inhibitors. Daily dependence on PPI's were eliminated in 75-80% of cases for up to six years in a 2014 study conducted by Testoni et al.. Although a TF procedure is not an option post bariatric surgery due to technical issues, it is available prior to LSG. With these surgeries working in tandem, patients may attain the benefits of both, as they are reciprocal in nature: TF provides anti-reflux barriers and LSG enables patients to lose weight, which ultimately decreases GER symptoms.

We propose that performing a TF procedure prior to a sleeve gastrectomy will result in a decrease in GERD symptoms similar to that of a LRYGB. In addition to evaluating symptoms, we will perform endoscopy screening post bariatric surgery at one, three, five and 10 years or more often as indicated , to assess for asymptomatic GERD and its sequelae..

Population to be Reviewed

1. Patient Identification

1. Patients seen for bariatric surgery consultation who report a history or current symptoms of GERD, or who are taking some form of medication for treatment of GERD, are asked to complete the Gastroesophageal Reflux Disease-Health Related Quality of Life Questionnaire .The GERD-HRQL is a validated, reliable and practical standard instrument which assesses the impact and severity of reflux symptoms on a patient's quality of life. The use of the GERD-HQRL for this purpose reflects a standard of care in the evaluation of any patient presenting with GERD symptoms.
2. The GERD-HRQL consists of 11 questions which focus on disease symptoms such as heartburn, difficulty swallowing, bloating, and pain, as well as the effect of these symptoms on daily life and an individual's satisfaction with their current condition. Symptoms are scored from 0 to 5, 0= no symptoms, 1= symptoms noticeable but not bothersome, 2= symptoms noticeable and bothersome but not every day, 3= symptoms bothersome every day, 4= symptoms affect daily activities, 5= symptoms are incapacitating, and unable to do activities. The summation of this score represents the severity and frequency of typical GERD symptoms. A score of 13 or higher on the GERD-HRQL warrants further diagnostic workup which may include the following: esophagogastroduodenoscopy, esophageal ambulatory pH study, esophageal manometry, and an upper gastrointestinal series.
3. Each patient is then presented at the GERD conference where treatment options are discussed and determined. The GERD conference is a multi-disciplinary meeting in which the patient's diagnostic results are presented in consideration of their personal history and comorbidities; based on these results, medical history and present status, treatment plans are discussed in order to provide the patient with the best possible outcome.
4. Treatment options are then presented to the patient, who ultimately decides the course of action. In general, patients are allowed to choose the surgical option that meets their treatment goals if they are able to demonstrate a clear understanding of the risks, benefits and indications for each choice. Therefore, patients are not randomized to one procedure.
5. GERD conferences will be retrospectively reviewed from March 2018 to February 2020 to identify bariatric patients with GERD who chose to undergo the TF procedure followed by the LGS or LRNGB. Thereafter, a continuing review following each GERD conference identifies patients suitable for study inclusion.
6. Patients who chose to undergo the TF to Sleeve route or who chose to undergo the LRYGB will be asked to consider consenting for their information to be part of this study. All patients who meet the proposal criteria will be approached by the study researchers until there are 60 patients enrolled in each category. Upon agreement, the patient's consent of the study will be appropriately documented.
7. Patients who choose LSG or TF to LSG will undergo screening endoscopies at the following postoperative LSG intervals: 12 months, three years, five years and 10 years.
8. A cohort of 60 patients who presented preoperatively with no evidence of GERD and underwent LSG, and who complete standard surveillance endoscopy postoperatively will be included in the study to provide a baseline from which to compare effectiveness of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bariatric patients who have documented GERD per GERD-HRQL at initial consultation and confirmed by preoperative testing
* 60 bariatric patients who received or plan to have the TF procedure prior to Sleeve Gastrectomy
* 60 bariatric patients who underwent or plan to undergo Roux-en-Y Gastric Bypass
* Male or female
* Ages 18 or older
* Bariatric patients who have no evidence of GERD per GERD-HRQL at initial consultation or on preoperative testing.
* 60 bariatric patients who received or plan to undergo LSG and who complete surveillance endoscopy one year postoperatively

Exclusion Criteria:

* Incomplete records missing any component of the demographic data to be analyzed
* Patients who undergo Roux-en-Y Gastric Bypass conversion from Sleeve Gastrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen for bariatric surgery consultation who report a history or current symptoms of GERD, or who are taking some form of medication for treatment of GERD, are asked to complete the Gastroesophageal Reflux Disease-Health Related Quality of Life Questionnaire GERD-HRQL. The GERD-HRQL is a validated, reliable and practical standard instrument which assesses the impact and severity of reflux symptoms on a patient's quality of life. The use of the GERD-HQRL for this purpose reflects a standard of care in the evaluation of any patient presenting with GERD symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2032-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure change in reflux symptoms, impact of symptoms, and satisfaction of current status with the Gastroesophageal Reflux Disease Health Related Quality of Life GERD HRQL-RSI Questionnaire | TS Cohort : Initial consultation, up to 6 weeks post fundoplication, up to 6 months post sleeve gastrectomy. RNY Cohort : At initial consultation, up to 6 months post RNY
  The GERD HRQL-RSI Questionnaire quantifies the symptoms of reflux the patient experiences, as well as the impact of symptoms on their daily life, and their satisfaction with their current status. The questionnaire also evaluates reflux medication use, which is another measure of treatment effectiveness. Items are rated on a scale of 0-5. The lowest possible score equals no symptoms.

SECONDARY OUTCOMES:
Measure change in Body Mass Index, BMI | TS Cohort: Initial Consultation, up to 6 weeks post fundoplication, up to 6 months post sleeve gastrectomy, 12 months post LSG. For the RNY Cohort, Initial Consultation and up to 6 months post RNY and 12 month post RNY.
  BMI is measured at initial consultation, up to 6 weeks post fundoplication, up to 6 months post LSG or RNY, and 12 months post LSG or RNY. It is a variable that may influence reflux symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Antonetti, MD, Principal Investigator — Lexington Health Incorporated
Locations (1):
- Lexington Health Incorporated, West Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, ICF
Time Frame: A date relative to the time when summary data are published.

REFERENCES:
- [Background] Barr AC, Frelich MJ, Bosler ME, Goldblatt MI, Gould JC. GERD and acid reduction medication use following gastric bypass and sleeve gastrectomy. Surg Endosc. 2017 Jan;31(1):410-415. doi: 10.1007/s00464-016-4989-4. Epub 2016 Jun 10. PMID 27287901
- [Background] DuPree CE, Blair K, Steele SR, Martin MJ. Laparoscopic sleeve gastrectomy in patients with preexisting gastroesophageal reflux disease : a national analysis. JAMA Surg. 2014 Apr;149(4):328-34. doi: 10.1001/jamasurg.2013.4323. PMID 24500799
- [Background] Rondelli F, Bugiantella W, Vedovati MC, Mariani E, Balzarotti Canger RC, Federici S, Guerra A, Boni M. Laparoscopic gastric bypass versus laparoscopic sleeve gastrectomy: A retrospective multicenter comparison between early and long-term post-operative outcomes. Int J Surg. 2017 Jan;37:36-41. doi: 10.1016/j.ijsu.2016.11.106. Epub 2016 Nov 29. PMID 27913235
- [Background] Tai CM, Huang CK. Increase in gastroesophageal reflux disease symptoms and erosive esophagitis 1 year after laparoscopic sleeve gastrectomy among obese adults. Surg Endosc. 2013 Oct;27(10):3937. doi: 10.1007/s00464-013-3022-4. Epub 2013 May 25. No abstract available. PMID 23708727
- [Background] Testoni PA, Testoni S, Mazzoleni G, Vailati C, Passaretti S. Long-term efficacy of transoral incisionless fundoplication with Esophyx (Tif 2.0) and factors affecting outcomes in GERD patients followed for up to 6 years: a prospective single-center study. Surg Endosc. 2015 Sep;29(9):2770-80. doi: 10.1007/s00464-014-4008-6. Epub 2014 Dec 6. PMID 25480624
- [Background] Trad KS, Turgeon DG, Deljkich E. Long-term outcomes after transoral incisionless fundoplication in patients with GERD and LPR symptoms. Surg Endosc. 2012 Mar;26(3):650-60. doi: 10.1007/s00464-011-1932-6. Epub 2011 Sep 30. PMID 21959689